CLINICAL TRIAL: NCT05325944
Title: Digital Mental Health Intervention for Nonsuicidal Self-Injury in Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH128410 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Nonsuicidal Self Injury; Suicidal Ideation; Depression; Anxiety
Keywords: Digital Mental Health; Nonsuicidal Self Injury; mHealth; Mobile phone; Smartphone; Coach; Conversational Agent
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-guided digital intervention for NSSI (Experimental): The self-guided digital intervention for NSSI will consist of 8 weekly modules containing psychoeducation and skill-based practice, and daily ecological momentary assessments. All content is delivered by a highly interactive conversational agent that guides users through the app content via a text-like interface.
  Interventions: Behavioral: Self-guided digital intervention for NSSI
- Digital intervention for NSSI with coaching (Experimental): The self-guided digital intervention for NSSI will consist of 8 weekly modules containing psychoeducation and skill-based practice, and daily ecological momentary assessments. All content is delivered by a highly interactive conversational agent that guides users through the app content via a text-like interface. This arm will additionally receive lightweight coaching which consists of a one 20-30 minute engagement call at the beginning of treatment. Thereafter, coaches will check in with participants via medium of participants choice twice per week and respond to patient texts, calls, or emails.
  Interventions: Behavioral: Digital intervention for NSSI with coaching
- Active control (Active Comparator): The active control arm will receive 8 weekly modules with psychoeducational components only, without the interaction features or EMA for personalization.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Self-guided digital intervention for NSSI — Psychoeducational content, skill-based practice, and daily ecological momentary assessments will be delivered over an 8-week period.
  Psychological strategies center on cognitive behavioral principles and acceptance-based emotional regulation strategies. Daily EMAs assess NSSI and use of cognitive, behavioral, and emotion regulatory strategies.
  Arms: Self-guided digital intervention for NSSI
Behavioral: Digital intervention for NSSI with coaching — Psychoeducational content and psychological strategies center on cognitive behavioral principles and acceptance-based emotional regulation strategies. Daily EMAs assess NSSI and use of cognitive, behavioral, and emotion regulatory strategies. Human coaching will be used to support intervention use and engagement twice per week via text, call or email.
  Arms: Digital intervention for NSSI with coaching
Behavioral: Active control — Psychoeducational content and psychological strategies center on cognitive behavioral principles and acceptance-based emotional regulation strategies.
  Arms: Active control

SUMMARY:
This is a feasibility trial of a digital mental health intervention aimed at young adults (ages 18-25) with nonsuicidal self-injury and who are not currently engaged in mental health treatment. We will pilot three arms: a self-guided DMHI, the DMHI with low-intensity coaching, or an active control which will involve the delivery of non-interactive psychoeducational content via the same app interface. The primary goals of this project are to evaluate the feasibility of the intervention and trial procedures in preparation for a fully-powered randomized-controlled trial.

DETAILED DESCRIPTION:
The primary purpose of this trial is to test the feasibility of conducting a randomized controlled trial (RCT) of an 8-week digital mental health intervention (DMHI) for non-treatment engaged young adults with repeated nonsuicidal self-injury. The DMHI will be a highly interactive conversational agent that conveys psychoeducational content and guides participants through skill-based activities. We will conduct a 3-arm feasibility trial, randomizing participants to receive the self-guided DMHI, the DMHI with low-intensity coaching, or an active control which will involve the delivery of non-interactive psychoeducational content via the same app interface. Initial randomization will be generated in permuted blocks of 6 using a computer program, with participants assigned on a 1:1:1 ratio. To prevent allocation bias, randomization will be conducted by the biostatistician, who will not inform the study team of the treatment arms until the baseline assessment has been completed and the patient has been enrolled. The control group will serve as the reference group to verify the effectiveness of the DMHI while the comparison of self-guided to coached deployments will evaluate the added benefit of coaching.

The primary clinical outcome measures will be frequency of NSSI behavior (ABASI) and frequency of NSSI urges (ABUSI). Secondary outcomes will include suicidal ideation (DSI-SS), depressive symptom severity (PHQ-9), and anxiety symptom severity (GAD-7).

This study will enroll individuals who have meet the following eligibility criteria: 1) current NSSI, defined as 2+ self-injury episodes (e.g., cutting, burning) in the past month; 2) Age 18 to 24; 3) English language skills sufficient to engage in the consent and intervention procedures. Participants will be excluded if they 1) Have a severe mental illness diagnosis (e.g., psychotic disorder); 2) Are imminently suicidal, with a plan and intent; or 3) Are currently receiving psychotherapy.

Coaching will consist of providing users with support and accountability via positive reinforcement, goal and expectation setting, and monitoring. Coaching outreach will focus on adherence to the treatment but will not provide treatment advice. Coaches will provide a brief (20-30 minute phone call or equivalent depending on the medium) engagement phone call. Thereafter, coaches will check in with participants via messaging, phone call, or email, twice per week and respond to patient messages.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-24 *The age to provide consent in Nebraska is 19. Individuals recruited from the state of Nebraska must be 19 or older.
* Current NSSI, defined as self-injury on 2 or more days in the past month
* Has a smartphone
* English language skills sufficient to engage in the consent and intervention procedures

Exclusion Criteria:

* Serious mental illness for which intervention would be contraindicated (e.g., psychotic disorder, manic episode, etc.)
* Severe suicidality (i.e., experiencing suicidal ideation with a plan and intent to act)
* Current engagement in psychotherapy

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Alexian Brothers Assessment of Self-Injury - Methods checklist | 16 weeks
  16-item checklist that assesses the frequency (days/times) of common NSSI methods within the past month.
Alexian Brothers Urges to Self-Injure Scale | 16 weeks
  5-item self-report measure assessing the intensity and frequency of NSSI urges. Higher scores mean more intense urges to self-injure. Minimum score: 0; maximum score: 30.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | 16 weeks
  10-item self-report measure assessing depression symptom severity. Higher scores mean greater symptom severity. Minimum score: 0; maximum score: 27.
Generalized Anxiety Disorder-7 | 16 weeks
  8-item self-report measure assessing generalized anxiety disorder symptom severity. Higher scores mean greater symptom severity. Minimum score: 0; maximum score: 21.
Borderline Evaluation of Severity Over Time | 16 weeks
  15-item self-report measure assessing borderline symptom severity. Higher scores mean greater symptom severity. Three domains: Thoughts and Feelings, Behaviors-Negative, Behaviors-Positive. Minimum score: 12; maximum score: 72.
Depression Symptom Inventory - Suicidality Subscale | 16 weeks
  4-item self-report questionnaire assessing the frequency and intensity of suicidal thoughts over previous two weeks. Higher scores signal greater frequency and severity of suicidal thoughts. Minimum score: 0; maximum score: 12.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylee C Kruzan, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through and managed by the NIMH Data Archive (NDA). De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of the primary outcome papers.
Access Criteria: The NIMH Data Archive is managed by the NIMH. Access criteria are determined by the NIMH.
URL: https://nda.nih.gov/